CLINICAL TRIAL: NCT06140641
Title: Effects of Supplementing the Bifidobacterium Longum BL21 on BMI, Metabolic Indicators, and Gut Microbiota in Overweight/Obese Adults: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Effects of the Bifidobacterium Longum BL21 on BMI, Metabolic Indicators, and Gut Microbiota in Overweight/Obese Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Hospital of Shandong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KYLL-202307-007
Record Dates: First submitted 2023-09-07; First posted 2023-11-20 (Actual); Last update posted 2023-11-20 (Actual); Status verified 2023-09

CONDITIONS: Overweight/Obese Adults
MeSH Terms: conditions — Overweight | interventions — Probiotics

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): Daily administration of placebo for 8 weeks.
  Interventions: Dietary Supplement: Probiotics
- Probiotics group (Experimental): Daily administration of Bifidobacterium Longum BL21 for 8 weeks.
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — Bifidobacterium Longum BL21 or placebo for 8 weeks.
  Other Names: Placebo

SUMMARY:
The goal of this study is to investigate the effects of Bifidobacterium longum subspecies BL21 on BMI, metabolic indicators, and changes in gut microenvironment microbiota in overweight/obese adults.

The blood, urine, and feces samples of the subjects need to be collected at 0,4 and 8 week and promptly tested in the laboratory. During the intervention period, all groups of subjects were required to take the corresponding products daily and record adverse reactions.

DETAILED DESCRIPTION:
The goal of this study is to investigate the effects of Bifidobacterium longum subspecies BL21 on BMI, metabolic indicators, and changes in gut microenvironment microbiota in overweight/obese adults. Randomized grouping was used to provide probiotic BL21 or placebo intervention. The total duration of the study is 8 weeks, including 8 weeks (1-8 weeks) of intervention expectations. The subjects were followed up at weeks 2 and 6, and sampled at weeks 0, 4, and 8. After the intervention during the follow-up period, blood, urine, and feces samples of the subjects need to be collected and promptly tested in the laboratory. During the intervention period, all groups of subjects were required to take the corresponding products daily and record adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) ≥ 24kg/m2 indicates overweight, and BMI ≥ 28kg/m2 indicates obesity;
2. Willing to take the test formulation daily during the study period;
3. Subjects who understand clinical research and commit to complying with research requirements and procedures.

Exclusion Criteria:

1. Patients with serious chronic diseases (heart, liver, kidney, hematopoietic system, tumor and other serious diseases, mental disease and organ surgery history, diabetes, etc.) and complications;
2. Patients with severe allergies and immune deficiencies;
3. Pregnant, breastfeeding, or expectant women during the study period
4. Patients with a clear history of gastrointestinal diseases (ulcers, irritable bowel syndrome, etc.);
5. Have a history of intervention with lipid-lowering drugs or health products within the past 2 months;
6. Individuals who have used antibiotics within the past two weeks;
7. Failure to consume the test sample as required, or failure to follow up on time, resulting in uncertain efficacy
8. Subjects deemed unsuitable by other researchers to participate.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2023-11-10 (Estimated); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Effects of intervention with Bifidobacterium longum BL21 on the gut microbiota in overweight/obese adults | 0, 4 and 8 week
  Take stool for microbial community sequencing

SECONDARY OUTCOMES:
Effects of intervention with Bifidobacterium longum BL21 on the BMI in overweight/obese adults. | 0, 4 and 8 week
  Record BMI

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhou, MD, Principal Investigator — Qilu Hospital of Shandong University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang X, Xing Z, Wang R, Zhang G, Liu G, Li Z, Li L. Multi-omics analyses the effect of Bifidobacterium longum subsp. longum BL21 supplementation on overweight and obese subjects: a randomized, double-blind, placebo-controlled study. Nutr Metab (Lond). 2025 Jul 17;22(1):79. doi: 10.1186/s12986-025-00969-2. PMID 40676704